CLINICAL TRIAL: NCT06774183
Title: Effect of Presbyopia Correction on Livelihood and Repayment Among Solar Customers in Western Region, Kenya: Evaluating the Impact of Providing Near Vision Correction to Solar Customers
Brief Title: Effect of Presbyopia Correction on Livelihood and Repayment Among Solar Customers in Western Region, Kenya
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dot Glasses Kenya (Other)
Collaborators: Queen's University, Belfast (Other); University of Stellenbosch (Other); Sun King (Unknown); Livelihood Impact Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P1751-2024
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Presbyopia Correction; Visual Impairment and Blindness (Excl Colour Blindness); Repayment Behaviour; Livelihoods
Keywords: Presbyopia; Near visual impairment; Near vision glasses; Income; Kenya; Rural
MeSH Terms: conditions — Vision Disorders; Blindness; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Near vision glasses (Experimental): Provision of NVGs for presbyopia correction at baseline for study duration
  Interventions: Other: Near vision glasses for presbyopia correction
- No glasses (No Intervention): Participants in the no intervention control group will be followed over the same period as the near vision glasses intervention group but will have no near vision glasses provided (glasses will be provided at the end of the study).

INTERVENTIONS:
Other: Near vision glasses for presbyopia correction — Provision of near vision glasses for presbyopia correction to individuals who did not previously have glasses and have correctable presbyopia
  Arms: Near vision glasses

SUMMARY:
With age, people lose the ability to see things that are near them clearly. This is known as presbyopia. Although this is a normal ageing process, it can be corrected with near vision eyeglasses - colloquially known as reading glasses - and people should not have to "put up with" poor near vision. By improving the ability to see things that are up-close, near vision eyeglasses allow people to perform tasks with greater ease. This improves their quality of life, and increases their productivity and income. DOT Glasses provides people in East Africa with a range of eyeglasses, including those to improve near vision.

In addition, products sold to communities through loans repaid at regular intervals (known as asset financing), allow people in underserved communities to harness electricity through solar products and to own electronic devices, such as mobile phones. This also improves their quality of life, and increases their productivity and income. Sun King is one of the leading providers of solar products through loans in Kenya.

This study will gather evidence and insights from existing Sun King customers with poor near vision in Busia, Siaya, Vihiga and Kakamega. The investigators will explore how much giving people glasses to improve their near vision impacts their ability to make repayments, their incomes and livelihoods, and their overall quality of life. It will also be studied how the glasses affect participants usage of the solar device or mobile phone.

DETAILED DESCRIPTION:
Aim:

To identify the impact on SHS and mobile phone use, repayment behaviour and income, of providing near vision glasses (NVGs) to customers with near vision impairment (NVI).

Primary objective:

● To determine the effect of presbyopia correction via NVGs, on SHS and mobile phone repayment behaviour:

* The proportion of total payments made on time
* Percentage of expected revenue collected within a six month time period

Secondary objectives:

* To determine the proportion of time SHS and mobile phones products are enabled among NVGs users
* To assess the effect of NVGs on quality of life among Solar Home System users.
* To measure the effect of NVGs on livelihood and income among Solar Home System users.
* To determine the value that Solar Home System users attached to the solar lighting and daily/weekly time using it.

POPULATION Sun King SHS or mobile phone (purchased on credit) users, aged 40 years or above, with presbyopia, who purchased their product at least 3 months ago and have at least 6 months of repayments remaining.

INTERVENTION Provision of NVGs for presbyopia correction.

CONTROL Delayed provision of NVGs, presbyopia correction.

TIME FRAME 6 months

HYPOTHESIS Correcting presbyopia with NVGs improves the rate of SHS or mobile phone repayments made on time.

NULL HYPOTHESIS Correcting presbyopia with NVGs does not change the rate of repayments made or the proportion of time the participants have their system enabled.

STUDY DESIGN Randomised Control Trial.

STUDY AREA The study area includes rural, peri-urban and urban communities in Busia, Siaya, Vihiga and Kakamega in Western Kenya

SAMPLE SIZE DETERMINATION Mean solar product repayments to Sun King for the entry level category, products priced between KES 7,000 and 30,000, are KES 405 per month. To be able to identify a 10% difference in repayments between the groups, with a two-sided significance level of p=0.05 and power of 90%, a sample size of 461 per group is required. The investigators will screen 1,480 people, of which it is expected 1085 to meet the enrolment criteria. 543 will be randomly allocated to join the experimental group who will be provided their glasses at the start of the study and 543 will be randomly allocated to join the control group who will receive their glasses at the end of the study. The investigators expect the attrition rate to be similar across both groups, at ~15%. This will give us a final sample per group of at least 461.

SAMPLING PROCEDURES A software application will be used to randomly select whether participants go into the study or control group. The application will randomly select from the participants list, then randomly invite participants on one of two days per locality for the screening, provision of NVGs and baseline surveys. The day attended will determine participants' allocation to the glasses or control groups.

All participants on day two will receive glasses and all on day one do not (control). Neither group will be informed beforehand if they are receiving glasses or not; they will only be invited for a screening.

* Glasses will not be dispensed on the first day at each location and then will be dispensed on the second day.
* When contacted, all participants will be invited for screening and told that they will receive eyeglasses at a date to be confirmed.

RECRUITMENT OF STUDY SUBJECTS

Sun King will call existing customers with the following criteria to invite them to participate in the study:

1. Aged over 40 years.
2. Purchased their product >=3 months ago and have >=6 months of repayments remaining on their PAYG contract.
3. The product is in the entry level category, priced between KES 7,000 and 30,000 (USD 46 and 196 at current exchange rates).
4. Reside in the counties of focus.

If they are willing to participate they will be asked if they have a pair of NVGs. If they do not have a pair, they will then be added to the initial participant list. If they have a pair, they will be excluded from selection. The selected study participants will be asked to complete and sign a consent form prior to the initial assessment and then randomly allocated to the experimental or control group.

Participants will receive compensation for travel expenses of 300 KSH

Data collection methodology

The data collection will be primarily quantitative. The data will be collected through:

1. Sun King's customer relationship management system, which records each client's product details, repayment schedule, payment details and the duration of the product's activation. This will be shared for analysis in a spreadsheet.
2. Individual surveys, using a semi-structured questionnaire. The surveys will be conducted in-person using Kobo Toolbox on mobile devices.
3. NVA test.

RESEARCH STAFF TRAINING

1. For the study the study team will be working with GMaurich Insights, a social research agency whose data scientists have over 20 years of combined experience.
2. GMaurich will provide Research Assistants (RAs) for the study.
3. DOT Glasses take the RAs through a 1-day training. The curriculum will cover:

   1. Research ethics and informed consent.
   2. Introduction to eye health and visual acuity.
   3. How to screen using the NVA chart.
   4. How to assess, at a basic level, if there may be more complicated eye conditions, and the referral process for other eye issues. It will be made clear to participants that this vision screening does not constitute a thorough ophthalmic examination, and that they should seek assessment for other visual/ocular symptoms elsewhere.
   5. How to distribute the glasses.
   6. Explaining to participants how to use the glasses and which tasks they should/should not be used for.
   7. Going through the question set.
4. GMaurich RAs will then need to pass a DOT Glasses practical assessment to be able to distribute the glasses.

DATA COLLECTION

1. A sample of 20 surveys will be completed to pilot the tool and stress-test the process.

2. Participants will be invited to a convenient location for the data collection. Depending on the day, the participants will be assigned to either the study or control group.

3. Data collection procedure in the field:

1. The RAs will explain the study purpose and process to the participant, and obtain written, informed consent before proceeding.
2. Conduct a DVA test with participants needing to achieve a minimum of 20/40.
3. Conduct a NVA test using Precision Vision Near Vision Chart:

i. Test presenting Near Visual Acuity. ii. Assess required near correction lens power (dioptres). iii. Retest corrected NVA. iv. Refer to a specialist if:

1. The participant has NVA worse than N6 at 40 centimetres and is not correctable by any of the available lenses.
2. The participant has other visible ocular pathology. d. Conduct the survey. e. For the study group: i. Provide the correct power and fit the glasses. ii. If no NVGs are required, offer sunglasses for their time and participation. f. For the control group: i. Assess the correct power, but delay glasses provision. ii. The eyeglasses will be provided at the end line.

4. Follow up period:

a. Intervention group: i. At 3 months participants will have an over the phone follow up to ask whether or not they are using the glasses.

ii. At 6 months follow up questionnaire and eye screening in person. b. Control group: i. At 6 months followed up questionnaire, eye screening and distribution of glasses.

COLLECTED DATA An overview of key question areas in the study tools is outlined below. Participant demographics

* Age
* Gender
* Location
* Education level
* Marital status
* Household size

Credit Questions

* Type of Pay-As-You-Go device they have?
* How and who pays for the device?
* Priority of paying for the device?

Solar questions

* Usage of product?
* Reasons for not paying?
* Vision challenges with the solar product?

Income and livelihoods

* Income sources and monthly income
* Income adequacy questions (perceived)

Vision-related quality of life assessment

● focusing on how their poor near vision has affected their daily lives.

At the end line, participants will be asked questions that measure their use of NVGs and the impact they have made on the above categories. With the control group getting a similar questions set.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years or older
* NVI secondary to presbyopia: presenting NVA <N6 at 40cm, correctable with NVGs to N6 or better at 40cm.
* Purchased their product >=3 months ago with >= 6 months of repayments remaining on their PAYG contract.
* The product is in the entry level category, priced between KES 7,000 and 30,000 (USD 46 and 196 at prevailing exchange rates during writing).
* Do not currently own a pair of NVGs.
* Living in a target counties of Busia, Siaya, Vihiga or Kakamega.

Exclusion Criteria:

* Age under 40 years.
* Distance Visual Acuity of worse than 20/40.
* Already own NVGs.
* Presenting NVA N6 or better at 40 centimetres.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1085 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Repayment behaviour - time | Measured at baseline and end of the study (6 months)
  The proportion of total payments made on time
Product usage | Measured at baseline and end of the study (6 months)
  The proportion of time solar home systems and mobile phones products are enabled
Repayment behaviour - percentage revenue | Measured at baseline and end of the study (6 months)
  Percentage of expected revenue collected by the solar home system provider within a six month time period

SECONDARY OUTCOMES:
Vision related quality of life | Measured at baseline and end of the study (6 months)
  Changes in perceived vision related quality of life assessed by questionnaire.
  Vision related quality of life will be assessed by 9 questions relating to how much difficulty the participant has in performing day to day tasks relating to their eyesight. Questions are answered on a scale from no difficulty at all to having to unable to perform the task due to eyesight issues.
Income | Measured at baseline and end of the study (6 months)
  Changes in self-reported income assessed by questionnaire.
  Participants will be asked how they generate an income and for each income source they will be asked how much they make per month from the income source (in KES).
Livelihood | Measured at baseline and end of the study (6 months)
  Changes in livelihood (source of income) assessed by questionnaire.
  Participants will be asked what there source of income is with the option to select multiple sources of income.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MEng, Principal Investigator — DOT Glasses

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised IPD data may be shared with other researchers for future research.

REFERENCES:
- [Background] Sehrin F, Jin L, Naher K, Das NC, Chan VF, Li DF, Bergson S, Gudwin E, Clarke M, Stephan T, Congdon N. The effect on income of providing near vision correction to workers in Bangladesh: The THRIVE (Tradespeople and Hand-workers Rural Initiative for a Vision-enhanced Economy) randomized controlled trial. PLoS One. 2024 Apr 3;19(4):e0296115. doi: 10.1371/journal.pone.0296115. eCollection 2024. PMID 38568883
- [Background] Reddy PA, Congdon N, MacKenzie G, Gogate P, Wen Q, Jan C, Clarke M, Kassalow J, Gudwin E, O'Neill C, Jin L, Tang J, Bassett K, Cherwek DH, Ali R. Effect of providing near glasses on productivity among rural Indian tea workers with presbyopia (PROSPER): a randomised trial. Lancet Glob Health. 2018 Sep;6(9):e1019-e1027. doi: 10.1016/S2214-109X(18)30329-2. Epub 2018 Jul 23. PMID 30049615